CLINICAL TRIAL: NCT06845917
Title: Personalized Digital Remote Monitoring for Elderly Patients: Multicentric RCT Study
Brief Title: Personalized Digital Remote Monitoring for Elderly Patients
Acronym: EPOCARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EPOCA U&I (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EPOCA-CT-2024-001
Record Dates: First submitted 2025-02-13; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Elderly Patients; Polypathology; Multiple Chronic Conditions
Keywords: Elderly; Hospitalization; Decompensation; Multiple chronic conditions; Remote monitoring
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: Multicentric Randomized controlled trial with two arms (intervention vs. control) for remote monitoring system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm: standard follow-up (No Intervention): Patients in the control group will receive standard medical care from their general practitioner or their geriatrician. In addition to the standard follow-up, they will be contacted for data collection purposes.
- Intervention arm: Patients followed by a Remote Monitoring System (Experimental)
  Interventions: Device: Remote Patient Monitoring system

INTERVENTIONS:
Device: Remote Patient Monitoring system — RMS consists of an initial assessment visit and system installation: A nurse trained by the EPOCA team will conduct a comprehensive assessment of the patient's needs during a home visit within 48 hours of enrollment. This includes collecting biometric measurements, socio-economic profile, and completing a questionnaire with the patient. The initial visit also includes a consultation with a physician. All the information is transmitted to a digital platform accordingly a personalized care plan (PCP) will be defined. The nurse installs a telemonitoring kit for the patient and gives them instructions on how to use it.
  The PCP manager will be responsible for implementing and overseeing the patient care plan, including informing the relevant stakeholders. Patients will be monitored via regular data feedback from the connected devices, the physician and the PCP manager. The PCP manager will treat any identified anomalies or abnormalities and implement the necessary changes on the PCP.
  Arms: Intervention arm: Patients followed by a Remote Monitoring System

SUMMARY:
Objective This clinical investigation aims to evaluate whether the EPOCA Remote Monitoring System (RMS) enhances care for elderly patients with multiple chronic conditions and reduces unplanned hospitalizations.

Key Research Questions

This study will assess:

* Unplanned Hospitalizations: Does EPOCA RMS reduce the total number of unplanned hospital days over 12 months?
* Quality of Life & Costs: What is the impact of EPOCA RMS on patients' quality of life and overall healthcare costs?
* Survival Rates: Does EPOCA RMS improve survival rates compared to standard care?

Participant Criteria

Participants must:

* Be 75 years or older with at least three chronic conditions.
* Have experienced a hospitalization or fall in the past year.
* Be randomly assigned to either the EPOCA RMS group or a control group receiving standard care.
* Be monitored for 12 months, with data collected at multiple time points.

Study Design

* Type: Multicenter, randomized controlled trial (RCT).
* Sites: Conducted across 8 hospitals in France.
* Duration: 12-month follow-up.
* Sample Size: 700 participants (350 per group).
* Intervention Group: Remote monitoring through the EPOCA RMS, integrating connected devices and medical coordination.
* Control Group: Standard care follow-up.

Expected Outcomes

* Reduced unplanned hospital stays and emergency visits.
* Improved quality of life and patient satisfaction.
* Comprehensive cost-effectiveness analysis and economic impact assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years,
* Three or more chronic pathologies (e.g., diabetes, heart disease, depression, cancer, respiratory failure, renal failure, dementia),
* Hospitalization or fall at least once in the previous year (Y-1),
* Recently discharged from the emergency department (within 24 hours),
* Patients, with or without caregivers, who accepted to participate and provided informed consent.

Exclusion Criteria:

* Patients discharged to or having been institutionalized in nursing homes (EHPAD),
* Patients enrolled in another clinical trial
* Suicidal or hetero-aggressive risk in a patient alone at home,
* Homeless patients,
* Patients protected by the following French legal measure: "sauvegarde de justice"

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Cumulative number of unplanned hospitalization days | Over 12 months

SECONDARY OUTCOMES:
Number of unplanned hospitalizations | Over 12 months
Change in quality of life from baseline using EQ-5D-5L scale | Initial, 6 and 12 months
  The instrument utilized was the EQ-5D-5L questionnaire, which comprises a self-reported health state description and a visual analogue scale (VAS). The EQ-5D-5L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problem, slight problems, moderate problems, severe problems, and extreme problems. Index scores range from -0.59 to 1; where 1 is the best possible health state. Negative values represent health states perceived as worse than dead, which is equal to 0.
Total number of days of hospitalizations for acute decompensation | Over 12 months
Survival and mortality proportion | At 12 months

OTHER OUTCOMES:
Number of hospitalizations | At 30 days
Number of emergency department visits | At 1 and 12 months
Number of patients referred to an EHPAD or USLD (long-term care facility) | At 12 months
Number of patients who require hospitalization at inclusion, including the days of hospitalization | At inclusion
The level of satisfaction with follow-ups using in-house specific survey | At 12 months
  The satisfaction of patients regarding their care pathway will be evaluated through the administration of a questionnaire developed by the research team. The survey will include questions pertaining to the patients' satisfaction with the telehealth experience, any equipment-related issues, concerns about privacy, the perceived impact of the telehealth intervention on their overall health, ability to stay healthier, and their understanding of their illness. Patients will be requested to provide a rating of their care on a Likert scale, with 10 representing the highest satisfaction rating and scores. The control group will complete the identical survey, substituting the term "telehealth" with "usual home care services."
Patient experience and perceived quality of care using Patient Assessment of Chronic Illness Care (PACIC) survey | At 6 months and 12 months
  Patient experience will be assessed at two time points (6 and 12 months) using the Patient Assessment of Chronic Illness Care (PACIC) survey. The PACIC tool consists of a 20-item patient report instrument that assesses a patient's receipt of clinical services and actions consistent with the Chronic Care Model (CCM). Respondents rate how often they experience the content described in each item during the past six months. Each item is scored on a five-point scale, ranging from one (no or never) to five (yes or always). Patients rate the care received from their primary health care team (not just their personal physician) for the chronic illness that they identified as most impacting their life.
Health services utilization - Economic evaluation through Budget Impact Analysis | At 12 months
  The economic evaluation will be a Budget Impact Analysis (BIA) of the intervention from both perspectives, societal and the NHI ("Assurance Maladie").
  Endpoints are :
  * Number of hospitalizations, length of stay and reason of admissions
  * Emergency room (ER) admissions
  * The number of consultations with the attending physician
  * Supportive care (physiotherapist, psychologist, sophrologist, etc.)
  * Home care visits
  * Transport services (taxi, VSL, ambulance, SAMU)
  * Nursing home care visits. For each questionnaire, the number of times the resource was consumed within the follow-up time was collected.
  For each patient, the total RU for 1 year will be estimated and expressed as yearly frequencies.
  RU will be valued by applying unit costs to RU in both arms and the difference between them will be estimated for all endpoints. Total cost per patient will be estimated for a 12-month duration of study.
Caregiver burnout, when present | At inclusion and 12 months
  Will be assessed using the Mini Zarit scale
Costs per patient | At 12 months
  Will be calculated by applying unit costs to resource use, estimating the average costs per patient over a 12-month period from societal and payer ("Assurance maladie") perspectives
Level of personalization based on GERS-model for care personnalisation | At 12 months
  The level of personalization will be described according to the care personnalisation model (GERS) - "Managing Singularity on a Large-Scale"

IPD SHARING:
Plan to Share IPD: No